CLINICAL TRIAL: NCT05629208
Title: A Randomized, Blinded, Placebo-Controlled, Phase 2a, Proof-of-Concept Study to Evaluate Efficacy, Safety, and Tolerability of GS-5718 in Participants With Cutaneous Lupus Erythematosus (CLE)
Brief Title: Study of Edecesertib in Participants With Cutaneous Lupus Erythematosus (CLE)
Acronym: COSMIC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-497-6486; 2022-501523-24 (Other: European Medicines Agency)
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Cutaneous Lupus Erythematosus (CLE)
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Edecesertib (Experimental): Participants will receive edecesertib 30 mg, once daily starting on Day 1 for up to 12 weeks.
  Interventions: Drug: Edecesertib
- Edecesertib Placebo (Placebo Comparator): Participants will receive edecesertib placebo, once daily starting on Day 1 for up to 12 weeks.
  Interventions: Drug: Edecesertib Placebo

INTERVENTIONS:
Drug: Edecesertib — Tablets administered orally
  Other Names: GS-5718
  Arms: Edecesertib
Drug: Edecesertib Placebo — Tablets administered orally
  Arms: Edecesertib Placebo

SUMMARY:
The goal of this clinical study is to test how edecesertib (formerly known as GS-5718) can be useful in treating Cutaneous Lupus Erythematosus (CLE) in participants with CLE. Information on what is happening in the body relating to CLE, how the body processes, is affected by and responds to the study drug, and any study drug side effects will also be collected in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Either fulfill European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) 2019 classification criteria for systemic lupus erythematosus (SLE) and/or have biopsy confirmed Cutaneous Lupus Erythematosus (CLE) at any time.
* Must have active CLE at screening and Day 1. Individuals with acute CLE (ACLE) must have involvement of 2 distinct body areas.
* Cutaneous Lupus Erythematosus Disease Area and Severity Index activity - A (CLASI-A) score (excluding alopecia) of ≥ 8 and CLASI-A erythema score of ≥ 4 during screening and on Day 1. Individuals with SLE must have Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score of ≥ 4 at screening.
* Presence of at least 1 representative lupus skin lesion amenable to punch biopsy and individual willingness to undergo skin punch biopsy at 2 time points.
* Must have documented prior intolerance or inadequate response at any time (per investigator judgement) to protocol-specified treatments.

  * Topical corticosteroids or topical calcineurin inhibitors.
  * Oral corticosteroids.
  * Any other nonbiologic standard-of-care therapy, including, but not limited to: chloroquine, quinacrine, hydroxychloroquine, azathioprine, mycophenolate mofetil (MMF), leflunomide, dapsone, or methotrexate (MTX).
* Individuals willing to comply with all study visits and assessments.

Key Exclusion Criteria:

* Individuals with only chilblains lupus, lupus panniculitis, lupus tumidus and/or localized acute CLE involving only 1 distinct body area at screening and Day 1.
* Have highly active SLE (including but not limited to lupus nephritis, neuropsychiatric SLE, and/or vasculitis).
* Presence of active skin conditions other than cutaneous lupus that may interfere with assessing lupus-specific skin lesion(s) (eg, psoriasis, and/or drug-induced lupus).
* Meet protocol-specified infection or lab criteria.

  * Any active infection that is clinically significant (per investigator judgment).
* Any history of clinically significant liver disease.
* Significant cardiovascular disease.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in Cutaneous Lupus Erythematosus Disease Area and Severity Index Activity (CLASI-A) Score at Week 12 | Baseline, Week 12
  The CLASI is a standardized, validated measure of cutaneous lupus disease activity and damage, widely used in clinical trials. CLASI consists of CLASI - activity (A) and - damage (D) measurements. CLASI-A scores range from 0 to 70, with higher scores indicating more severe disease activity.

SECONDARY OUTCOMES:
Proportion of Participants With Cutaneous Lupus Activity Investigator Global Assessment (CLA-IGA) Score of 0 or 1 at Week 12 | Week 12
  The CLA-IGA is a measure of cutaneous lupus erythematosus (CLE) activity and will be recorded on a scale of 0 to 4, with 0 indicating "clear" and 4 indicating "severe".
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | First dose date up to 12 weeks plus 30 days
Percentage of Participants Experiencing Serious Treatment-emergent Adverse Events (TESAEs) | First dose date up to 12 weeks plus 30 days
Percentage of Participants Experiencing Laboratory Abnormalities | First dose date up to 12 weeks plus 30 days
Plasma Concentration of Edecesertib | Postdose at Week 2, Predose at Week 4 and 12, and Week 8 (anytime of the day)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (17):
- United States (12):
  - ARENSIA Exploratory Medicine, LLC, Phoenix, Arizona
  - Center for Dermatology Clinical Research Inc., Fremont, California
  - University of Colorado, Barbara Davis Center, Center for Clinical Research, Aurora, Colorado
  - Yale Center for Clinical Investigation (YCCI), New Haven, Connecticut
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Reliant Medical Research, Miami, Florida
  - HMD Research LLC, Orlando, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Dept. of Dermatology, Hospital of the University of Pennsylvania, Perelman Center for Advanced Medicine (PCAM), Philadelphia, Pennsylvania
  - Gulf Bank Medical Center, Houston, Texas
  - Clinical Investigations of Texas, Plano, Texas
- Germany (3):
  - Universitätsklinikum Carl Gustav Carus Klinik und Poliklinik für Dermatologie, Dresden
  - Universitatsklinikum Freiburg Klinik fur Dermatologie und Venerologie, Freiburg im Breisgau
  - Universitätsklinikum Leipzig AöR Klinik und Poliklinik für Dermatologie, Venerologie und Allergologie Klinische Forschungseinheit (KFE) - Haus 10, Leipzig
- Spain (2):
  - Hospital General de Granollers, Granollers
  - Hospital Universitario de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-497-6486